CLINICAL TRIAL: NCT01932541
Title: Open-Label Study of Latuda for the Treatment of Mania in Children and Adolescents 6-17 Years Old With Bipolar I, Bipolar II and Bipolar Spectrum Disorder
Brief Title: Open-Label Study of Latuda for the Treatment of Mania in Children and Adolescents 6-17 Years Old
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: On hold due to competing departmental studies
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Associate Professor of Psychiatry, Harvard Medical School; Director, Pediatric Bipolar Clinical and Research Program in Pediatric Psychopharmacology, Massachusetts General Hospital., Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-P-001524
Record Dates: First submitted 2013-08-20; First posted 2013-08-30 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Mania; Bipolar I; Bipolar II; Bipolar Spectrum Disorder; Bipolar Disorder
Keywords: Bipolar Disorder; Mania; Bipolar I; Bipolar II; Bipolar Spectrum Disorder; Pediatric
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latuda (Lurasidone) (Experimental)
  Interventions: Drug: Latuda (Lurasidone)

INTERVENTIONS:
Drug: Latuda (Lurasidone) — Latuda® (lurasidone) tablets taken by mouth once daily, between 20 mg and 120 mg a day.
  Other Names: Lurasidone; Latuda

SUMMARY:
This study is an 8-week open-label trial testing Lurasidone (Latuda®) as a treatment for mania in children and adolescents with Bipolar I, Bipolar II, and Bipolar Spectrum disorders. We hypothesize that Lurasidone will be safe, tolerable, and effective in improving the core symptoms of bipolar disorders in children and adolescents ages 6-17.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 6-17 years of age
2. Subjects must weigh at least 20 kg
3. Subjects with the diagnosis of bipolar I, bipolar II, or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features), by DSM-IV (Diagnostic and Statistical Manual IV), as manifested in clinical evaluation and/or the Mania module of the structured interview, completed by the study clinician. Bipolar Spectrum Disorder (or sub-threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but displays fewer elements in Criteria B (only require 2 items for elation category and 3 for irritability)
4. Subjects must score ≥ 20 on the YMRS (Young Mania Rating Scale)
5. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
6. Subjects and their legal representative must be considered reliable reporters.
7. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document (if ≥ 7 years old).
8. Subject must be able to participate in mandatory blood draws.
9. Subject must be able to swallow pills.
10. Subjects with co-morbid PDD (Pervasive Developmental Disorder) and depressive disorders will be allowed to participate in the study provided they do not meet any of the exclusionary criteria.
11. For concomitant therapy used to treat ADHD (Attention Deficit Hyperactivity Disorder), subjects must have been on a stable dose of the medication for 1 month prior to study enrollment, and the dose of the ADHD therapy cannot change throughout the duration of the study.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Uncorrected hypothyroidism or hyperthyroidism.
4. Non-febrile seizures without a clear and resolved etiology.
5. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months.
6. Judged clinically to be at serious suicidal risk or have a C-SSRS (Columbia Suicide Severity Rating Scale) score ≥ 4.
7. Any other concomitant medication with primary central nervous system activity other than specified in the Concomitant Medication portion of the Protocol.
8. Current diagnosis of schizophrenia.
9. Mental retardation (IQ < 75)
10. Pregnant or nursing females
11. Known hypersensitivity to Latuda®
12. A non-responder or history of intolerance to Latuda®, after treatment at adequate doses as determined by the clinician.
13. Severe allergies or multiple adverse drug reactions.
14. Subjects with a hematological disorder.
15. Subjects with diabetes.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale | Change from baseline at 12 weeks
  This is a widely used instrument that assesses symptoms of mania in clinical trials of adult and pediatric subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, M.D., Principal Investigator — Massachusetts General Hospital Clinical and Research Program in Pediatric Psychopharmacology
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States